CLINICAL TRIAL: NCT02425670
Title: Intravenous Autologous Bone Marrow-derived Stem Cells Therapy for Patients With Acute Ischemic Stroke: A Multi-Institutional Project
Brief Title: Stem Cell Therapy For Acute Ischemic Stroke Patients
Acronym: InVeST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: All India Institute of Medical Sciences (Other)
Collaborators: Ministry of Science and Technology, India (Other Government); Army Hospital Research And Referral, India (Other); Armed Forces Medical College, Pune (Other); Post Graduate Institute of Medical Education and Research, Chandigarh (Other); Sanjay Gandhi Postgraduate Institute of Medical Sciences (Other Government)
Responsible Party: Principal Investigator, Kameshwar Prasad, Professor and Head, Department of Neurology, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BT/pr6815/MED/14/880/2005AIIMS; REFCTRI000046, 19.04.2008 (Other: WHO)
Record Dates: First submitted 2015-04-07; First posted 2015-04-24 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2015-04

CONDITIONS: Middle Cerebral Artery Infarction; Anterior Cerebral Artery Infarction
Keywords: Brain attack; stroke; Ischemic stroke; stem cell therapy
MeSH Terms: conditions — Infarction, Middle Cerebral Artery; Infarction, Anterior Cerebral Artery; Stroke; Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bone marrow derived stem cells (BMSCs) (Experimental): BMSCs 30-500 million plus conventional management
  Interventions: Other: BMSCs
- Control (No Intervention): Control: conventional management

INTERVENTIONS:
Other: BMSCs — 30-500 million Autologous BMSCs will be given intravenously to patients with acute ischemic stroke (onset from 7 to less than 30 days).
  Other Names: Stem cell arm
  Arms: Bone marrow derived stem cells (BMSCs)

SUMMARY:
The purpose of this study is to determine whether patients with subacute ischemic stroke will benefit from infusion of patient's own bone marrow derived stem cells.

Primary Hypothesis: Intravenous injection of bone marrow mononuclear cells at a dose of 30 to 500 million in patients with subacute ischemic stroke results in reduction of infarct volume and improvement of neurological function compared to those without the injection.

Secondary Hypothesis: Patients receiving more than 100 million Bone marrow derived stem cells (BMSC) will have better outcome than those receiving fewer dosages of cells.

DETAILED DESCRIPTION:
Background: Stroke accounts for significant disability and there is need for novel treatment modality which can improve the functional outcome. In this randomized clinical trial, investigators proposed to examine stem cell therapy as a potential therapeutic modality. Stem cells in animal stroke models have shown reduction in infarct size and improvement in neurological function. Only one human clinical trial with intravenous autologous marrow stromal cell therapy of five patients has shown some benefit. The primary objective of this phase II study was to explore if there is favourable risk to benefit ratio for autologous bone marrow derived mononuclear stem cell therapy (BMSCs) in patients with acute ischemic stroke to justify a larger phase III trial.

Methods & Design: The study recruited 120 men and women aged 18-70 years presenting with acute ischemic stroke (7-29 days) and a NIHSS score of ≥ 7 and BI ≤ 50. Following baseline assessment (MRI Brain, Whole Body PET scan, EEG brain, CT scan Brain and clinical examination including National Institute of Health Stroke Scale (NIHSS), Barthel Index (BI), modified Rankin Scale (mRS), Glasgow Come Scale (GCS), participants were randomly allocated to two groups: conventional management alone (control group); or conventional management and autologous intravenous BMSCs transplantation (experimental group). Bone marrow was aspirated under local anaesthesia and the isolated BMSCs cells injected intravenously within 4 hours. The patients were monitored with hemogram & renal/liver function tests, CT scan brain at 36 hrs and clinical examination for a week. The patients were followed up to one year with periodic MRI brain at 3 months, 6 months, EEG & PET scan at 6 months and 1 year. The primary efficacy outcomes were difference between the two groups in the Modified Barthel index score and modified Rankin Scale score at six-month post-randomisation. The secondary efficacy outcomes are: NIHSS score at six-months and 1 year post-randomisation; and the modified Rankin scale score at 3 months and one year post-randomization, and functional status measured by barthel index (in binary scale <60 or >60 ) at six months and one year post-randomization. Dose response analysis were done by comparing outcomes in patients receiving various doses of bone marrow mononuclear cells.

Discussion: This phase 2 study was aimed to explore if there is a favourable risk-to-benefit ratio for stem cell therapy in patients with acute ischemic stroke. Investigators also planned to examine whether there is justification for phase III trial of autologous bone marrow derived mononuclear stem cell therapy for acute ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

Patients will be judged eligible if they have all of the following:

1. Sudden onset of focal neurologic deficit or impairment of consciousness,
2. Computerized tomographic or MRI scan of the head showing no primary haematoma, and relevant lesions within the Middle Cerebral Artery (MCA) and anterior cerebral artery (ACA) territory. Hemorrhagic changes in infarct are acceptable.
3. Age between 18 and 75 years
4. Seven days or more but less than 30 days since the onset of the qualifying event,
5. Glasgow Coma Scale score of above 8 at the time of randomization, in aphasic Eye and Motor score of more than 6,
6. Modified Barthel index score of 50 or less at the time of randomization.
7. NIHSS score of 7 or more points and inability to walk unaided or raise upper limb by 90 °
8. Patient is stable: A patient will be defined as stable when he has normal respiration, is afebrile, has BP less than mean arterial pressure of 125mm Hg (but no hypotension defined as systolic BP <90mmHg), has fasting venous blood sugar level less than 200mg % and normal urea/electrolytes for at least 48 hours.

Exclusion Criteria:

Patients meeting the inclusion criteria will be considered ineligible for the study if they have any one of the following:

1. Lacunar syndrome
2. Intubation
3. Posterior Circulation Stroke
4. Co-morbidity likely to limit survival to less than three years e.g. malignant diseases, hepatic or renal failure
5. Pre-stroke disability leading to dependence on others for activities of daily living,
6. Inaccessibility for follow-up
7. Allergy to local anaesthetic
8. Unwillingness to provide written informed consent by self or assent by next of kin.
9. Symptom of Acute myocardial infarction or acute involvement of any other organ.
10. Pregnancy
11. Human immunodeficiency virus (HIV)/hepatitis C virus (HCV)/HbsAg positive.
12. Patient is a part of any other trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2009-01; Primary Completion 2010-10 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Functional ability to perform activities of daily living on Modified Barthel Index Score | 6 months

SECONDARY OUTCOMES:
Neurological deficit on NIHSS score | 6 months and 1 year
Measurement of disability on Modified Rankin Scale | 3 months, 6 months and one year
Functional ability to perform activities of daily living on Modified Barthel Index (Functional status) on binary scale as independent (Barthel index > 60) or dead or dependent (Barthel Index <60) | 6 months and one year

CONTACTS AND LOCATIONS:
Overall Officials: Kameshwar Prasad, MBBS, MD, Principal Investigator — All India Institute of Medical Sciences
Locations (5):
- India (5):
  - Postgraduate Institute of Medical Education & Research, Chandigarh, Chandigarh
  - Armed Forces Medical College, Pune, Maharashtra
  - Army Hospital (Referral and Research Centre),, Delhi Cantonment, National Capital Territory of Delhi
  - All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi
  - Sanjay Gandhi Postgraduate Institute of Medical Sciences, Lucknow, Uttar Pradesh

REFERENCES:
- [Result] Prasad K, Sharma A, Garg A, Mohanty S, Bhatnagar S, Johri S, Singh KK, Nair V, Sarkar RS, Gorthi SP, Hassan KM, Prabhakar S, Marwaha N, Khandelwal N, Misra UK, Kalita J, Nityanand S; InveST Study Group. Intravenous autologous bone marrow mononuclear stem cell therapy for ischemic stroke: a multicentric, randomized trial. Stroke. 2014 Dec;45(12):3618-24. doi: 10.1161/STROKEAHA.114.007028. Epub 2014 Nov 6. PMID 25378424
- See also: link for published manuscript — http://stroke.ahajournals.org/content/45/12/3618.long